CLINICAL TRIAL: NCT05248776
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study to Evaluate Efficacy, Safety and Pharmacokinetics After 2-weeks Administration of CPL207280 (GPR40 Agonist) in Subjects With Type 2 Diabetes (T2D)
Brief Title: Efficacy, Safety and Pharmacokinetics Study of CPL207280 After 2-weeks Administration in Subjects With Type 2 Diabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Celon Pharma SA (Industry)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02GPR2021
Record Dates: First submitted 2022-02-04; First posted 2022-02-21 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — CPL207280

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo- controlled, parallel-group study to explore the efficacy, safety, tolerability and PK of 4 different doses of CPL207280 administered for 14 days orally.
Who Masked: Participant, Investigator
Masking Description: Double- Blind. The identity of IMP and placebo will not be known to investigators, research staff and participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CPL207280 60 mg (Experimental): 16 participants are to receive IMP at dose 60 mg.IMP will be administered for 14 days, every morning, after a minimum 8-hours overnight fast. Participants are to be randomized.
  Interventions: Drug: CPL207280
- CPL207280 120 mg (Experimental): 16 participants are to receive IMP at dose 120 mg. IMP will be administered for 14 days, every morning, after a minimum 8-hours overnight fast. Participants are to be randomized.
  Interventions: Drug: CPL207280
- CPL207280 240 mg (Experimental): 16 participants are to receive IMP at dose 240 mg. IMP will be administered for 14 days, every morning, after a minimum 8-hours overnight fast. Participants are to be randomized.
  Interventions: Drug: CPL207280
- CPL207280 480 mg (Experimental): 16 participants are to receive IMP at dose 480 mg. IMP will be administered for 14 days, every morning, after a minimum 8-hours overnight fast. Participants are to be randomized
  Interventions: Drug: CPL207280
- Placebo (Placebo Comparator): 16 participants are to receive masking placebo tablets once daily for 14 days, every morning, after a minimum 8-hours overnight fast. Participants are to be randomized
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CPL207280 — IMP is a tablet with CPL207280 as an Active Pharmaceutical Ingredient (API).
  Arms: CPL207280 120 mg; CPL207280 240 mg; CPL207280 480 mg; CPL207280 60 mg
Drug: Placebo — Matching placebo tablet.
  Arms: Placebo

SUMMARY:
The planned study is to evaluate the efficacy, safety and pharmacokinetic (PK) properties of CPL207280 after multiple (14 days) administration in patients with type 2 diabetes.

DETAILED DESCRIPTION:
A double-blind, randomized, placebo-controlled, parallel-group study of 4 different doses of CPL207280 administered orally for 14 days. Approximately 80 participants will be randomized at a 1:1:1:1:1 ratio to 5 arms to receive Investigational Medicinal Product (IMP) or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participant with type 2 diabetes who are newly diagnosed (no longer than 3 years before the study) managed with diet and exercise alone, or who failed to achieve adequate glycemic control on a stable dose of metformin and willing to discontinue it at least 10 days prior to randomization and during the study.
* Participant has fasting plasma glucose level less than or equal 180 mg/dL.
* Participant has calculated homeostasis model assessment for insulin resistance (HOMA-IR) value less than or equal to 7.
* Participant has body-mass index (BMI): ≥ 18.50 kg/m² and ≤ 40.00 kg/m².
* Participant should have a HbA1c concentration greater than or equal to 6.0% and less than or equal to 8.0%.
* Participant has not received treatment with weight-loss drugs within the 3 months prior to the study
* Participant has a systolic blood pressure less than or equal to 160 mm Hg and a diastolic blood pressure of less than or equal to 100 mm Hg.
* Participant has the clinical laboratory evaluations [including fasting clinical chemistry, hematology and complete urinalysis (excluding glucose results)] within the reference range for the testing laboratory, unless the investigator deems the out-of-range results to be not clinically significant.
* Participant has negative test results for hepatitis B surface antigen and antibody to hepatitis C virus, negative RT-PCR test results for COVID-19, negative antibody to HIV virus and no known history of human immunodeficiency virus.
* Participant is considered by the investigator to be in a good health (other than being diabetic) as determined during the medical history review, physical examination findings, electrocardiogram and vital sign results, and clinical laboratory evaluations.
* Participant has estimated Glomerular Filtration Rate (eGFR) greater than 60 mL/min/1.73m^2.
* A female is eligible to participate if she is not pregnant (negative serum pregnancy test ), not breastfeeding,
* Male participants must agree to use a barrier method of contraceptive during the study and for at least 90 days after the last dose of the study drug
* Participant has the ability and willingness to comply with the requirements and restrictions of the study protocol.

Exclusion Criteria:

* Participant has a c-peptide value less than 0.5 nmol/l.
* Participant has a history of abdominal surgery (except laparoscopic cholecystectomy or uncomplicated appendectomy), thoracic, or non-peripheral vascular surgery within 6 months prior to the study.
* Participant has a history of cardiac arrhythmia, systolic dysfunction, congestive heart failure, angina, myocardial ischemia or infarction, or stroke within 1 year prior to the study, or the presence of an abnormal ECG that, in the investigator's opinion, is clinically significant.
* Participant has a history of drug abuse or a history of alcohol abuse within 2 years prior to the study.
* Participant has a history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug. This criterion does not apply to basal cell or stage I squamous cell carcinoma of the skin.
* Participant has an alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase level above normal range for the testing laboratory, active liver disease.
* Participant has a total bilirubin greater or equal 2 mg/dL.
* Participant is/ was lifetime on any insulin treatment or takes other diabetes treatment (except metformin).
* Participant has a history of proteinuria ≥300 mg/day on a 12- or 24-hour urine collection within last year or an albumin/creatinine ratio greater or equal 300 μg/mg.
* Participant has a history of any clinically significant retinopathy, which is defined as more than moderate nonproliferative diabetic retinopathy, any stage of proliferative diabetic retinopathy or any history of laser-treated retinopathy.
* Participant has clinically significant peripheral or autonomic neuropathy.
* Participant has a lifetime history of ulcerative colitis or Crohn's disease, or has undergone gastric resection.
* Participant has a history of a psychiatric disorder that, in Principal Investigator opinion, will affect the subject ability to participate in the study.
* Participant has a lifetime history of angioedema.
* Participant has an acute, clinically significant illness within 30 days prior to the study or any other condition or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study.
* Participant is not able to comply with the study scheduled visits.
* Participant is participating in another investigational study or has taken any investigational drug within 90 days prior to the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy in lowering plasma glucose during the Oral Glucose Tolerance Test (OGTT) after 2 weeks of CPL207280 treatment | Day -2 and Day -14
  Change in plasma glucose, evaluated through area under the plasma glucose concentration- time curve AUC (0-3 h) during the OGTT.

SECONDARY OUTCOMES:
Change in plasma glucose maximal concentration (Cmax) level during the OGTT | Day -2 and Day 14
Change in plasma glucose concentration level at 2 hours timepoint level during the OGTT | Day -2 and Day -14
Change in Fasting Plasma Glucose (FPG) | Day 1 and Day 15
Change in Fasting Plasma Insulin (FPI) | Day 1 and Day 15
Change in Fasting Plasma Proinsulin | Day 1 and Day 15
Change in Fasting Plasma c-peptide | Day 1 and Day 15
Change in Fasting Plasma Glucagon | Day 1 and Day 15
Change in plasma insulin, evaluated through area under the plasma insulin concentration-time curve (AUC0-3 hours) during the OGTT | Day -2 and Day 14
Change in plasma insulin maximal concentration (Cmax) level during the OGTT | Day -2 and Day 14
Change in plasma insulin concentration at 2 hours time point plasma level during the OGTT | Day -2 and Day 14
Change in HbA1c value after 14 days of CPL207280 treatment | Day -14 and Day 15
Absolute change in homeostasis model assessment of ß-cell function (HOMA-ß) | Day -2 and Day 14
Number of Participants who experienced at least once Adverse Event related to the study product | Up to 28 days
Number of Participants who experienced at least once Hypoglycaemia episode | Up to 15 days
Number of Participants who discontinued study due to an Adverse Event related to the IMP | Up to 15 days
Number of Participants with abnormal laboratory values | Up to 15 days
Number of Participants with abnormal ECG values | Up to 15 days
Change from pre dose value to mean of post dose values of Total Bile Acids on Day 1 and 14 | Pre dose Day 1, Day 14, post dose Day 1, Day 14
CPL207280 maximum observed concentration (Cmax) | Day 1, Day 8, Day 14
CPL207280 time corresponding to occurence of Cmax (tmax) | Day 1,Day 8, Day 14
CPL207280 AUC from time zero to infinity (AUC 0-inf) | Day 1, Day 8, Day 14
CPL207280 apparent terminal elimination half-life (t1/2) | Day 1, Day 8, Day 14
CPL207280 apparent clearance (CL/F) | Day 1, Day 8, Day 14
CPL207280 apparent volume of distribution during terminal phase (Vz/F) | Day 1, Day 8, Day 14
CPL207280 concentration immediately prior to dosing (Ctrough) | Day 1, Day 8, Day 14,

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Jonak, Principal Investigator — BioResearch Group Sp. Z o.o.
Locations (1):
- BioResearch, Kajetany, Nadarzyn, Poland

IPD SHARING:
Plan to Share IPD: No